CLINICAL TRIAL: NCT04095702
Title: A Pilot Study to Look at the Use of Stabilizing (Weighted) Pacifier vs. the Use of a Traditional Non-Stabilizing (Non-Weighted) Pacifier to Improve Infant Comfort, Caregiver Satisfaction, and Safety During Non-Nutritive Sucking
Brief Title: Weighted Pacifier Vs. Non-Weighted Pacifier
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Englewood Hospital and Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E-19-782
Record Dates: First submitted 2019-08-22; First posted 2019-09-19 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Non-nutritive Sucking

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Weighted Pacifier (Experimental): Patient will receive a weighted pacifier for 48 hours of their stay in the NICU.
  Interventions: Other: Weighted Pacifier
- Non-Weighted Pacifier (Placebo Comparator): Patient will receive a standard non-weighted pacifier for 48 hours of their stay in the NICU.
  Interventions: Other: Non-Weighted Pacifier

INTERVENTIONS:
Other: Weighted Pacifier — The weighted pacifier is a standard of care pacifier with a weighted, breathable star attachment to help keep the pacifier from popping out of the neonates mouth during non-nutritive suck.
  Arms: Weighted Pacifier
Other: Non-Weighted Pacifier — The non-weighted pacifier is a standard of care pacifier that a neonate would receive if they were not part of this study.
  Arms: Non-Weighted Pacifier

SUMMARY:
This study will determine if it is beneficial to use a weighted pacifier in neonates.

DETAILED DESCRIPTION:
RCI-Pacifiers have been utilized for decades in the NICU to provide benifical Non-Nutritive Suck. They have been instrumental in transitioning premature infants from gavage to breast feeding Yiallouerou, S, et al, studied the effects of dummy/pacifier on autonomic activity during sleep and found pacifier use to be protective during sleep. Risks and Benefits of Pacifiers have cleary been identified Sexton, S and Natsale, R have identified that nonnutritive suck is a natural reflex for a fetus and newborn. Traditionally, the pacifier has been used as a method for fulfilling an infants innate desire to suckle. Study subjects will be introduced to either a standard/traditional pacifier (without stabilizing/weighted attachment) or a stabilizing/weighted pacifier. Standard/traditional pacifiers will be issued to patients that have been assigned an odd number study identifier and , stabilzing/weighted pacifiers will be issued to patients that have been assigned an even number study identifier. All eligible infants born at 30 weeks to 37.6 weeks who meet study criteria will be included. All staff/caregivers will be trained in proper placement of a stabilizing pacifier prior to use. Stabilizing pacifiers will not be placed on the infants chest. Traditional pacifiers will be used as standard of care at EH. The Neonatal Infant Pain Score (NIPS) scale and a caregiver survey will be used to determine efficacy.

ELIGIBILITY:
Inclusion

* 30 week-37.6 gestational age
* Patient is admitted to the NICU
* The patient has the ability to suck as noted in the patient's infant assessment flow sheet prior to enrollment

Exclusion

* Patient with an oral pharyngeal defect
* Patient with an oral feeding tube
* Patient with any medical reason that deems them unfit for the study as '''''''determined by the neonatologist
* Patient with sustained apnea during sucking

Ages: 30 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2021-11-18 (Actual)

PRIMARY OUTCOMES:
Safety determined by a Neonatal Infant Pain Scale (NIPS) score | 48 hours
  To determine if the weighted pacifier is safe in supporting non-nutritive suck. Neonates will be measured in facial expression, cry, breathing pattern, and state of arousal. Each category get a rating of 0 or 1, with 0 being negative and 1 being positive.
efficiency determined by an Efficiency of Loss scale | 48 hours
  To determine if the weighted pacifier is efficient in supporting non-nutritive suck. The neonates will be observed for a period of 10 minutes each time the pacifier is introduced. The observer will count the amount of time the neonate's pacifier pop from his/her mouth.

SECONDARY OUTCOMES:
Stress/ Discomfort determined by a Likert Scale | 48 hours
  To determine if a stabilized pacifier reduces infant stress/discomfort
Caregiver stress determined by a Likert Scale | 48 hours
  To determine if a caregiver's stress level decreases when an infant is provided with a stabilizing/weighted pacifier versus a traditional pacifier. The scale will consist of questions asking about the caregiver's stress. The caregiver will answer the questions with a 1-5 rating, with 1 being strongly disagree and 5 being strongly agree.

CONTACTS AND LOCATIONS:
Locations (1):
- Englewood Health, Englewood, New Jersey, United States